CLINICAL TRIAL: NCT03799497
Title: Neural Correlates of Self Body-shape Recognition in Anorexia Nervosa, an fMRI Activation Study
Brief Title: Neural Correlates of Self Body-shape Recognition in Anorexia Nervosa Mental
Acronym: Explorexie
Status: Completed | Type: Observational
Sponsor: University Hospital, Lille (Other)
Responsible Party: Sponsor
Other Study IDs: 2009_48; 2010-A00545-34 (Other: ID-RCB number, ANSM)
Record Dates: First submitted 2019-01-03; First posted 2019-01-10 (Actual); Last update posted 2020-09-16 (Actual); Status verified 2020-09

CONDITIONS: Anorexia Nervosa
Keywords: Anorexia nervosa; functional MRI (fMRI); self body-shape recognition
MeSH Terms: conditions — Anorexia Nervosa

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Patients suffering from Anorexia Nervosa: Subjects with a diagnostic of anorexia nervosa disorder
- Control group: Healthy subjects with no psychiatric disorder

SUMMARY:
Body Image distortion is a key diagnostic feature for Anorexia Nervosa. Patients suffering from Anorexia Nervosa tend to perceive themselves as fatter than they are. This bias might be at the origin of a reinforcement of anorectic behavior which might alter medical care. The objective of this study is to identify neural correlates of self-recognition in Anorexia Nervosa. Patients are hypothesized to activate the self-recognition network when seeing images of a fatter body shape than their own.

DETAILED DESCRIPTION:
Patients suffering from Anorexia Nervosa and control subjects (matched by age and study level) are recruited in medical care facilities in Lille's Metropolis. They are asked to identify their body shape when being presented with 3 different stimuli, i.e.real (RBS), estimated (EBS) and neutral body shape (NBS), in a functional magnetic resonance imaging or functional MRI (fMRI) machine. While answering to this identification paradigm, we hoped to identify modifications in the self body-recognition network.

ELIGIBILITY:
Inclusion Criteria:

* Providing informed, dated and signed consent (for minors, consent must be signed by both parents)
* With medical insurance
* With normal vision
* Only for the AN Group : Diagnosis of Anorexia Nervosa (AN) restrictive for at least one year and with a Body Masse index (BMI) between 14 and 18
* Only for the control Group : BMI between 18 and 25 and without any psychiatric disorder

Exclusion Criteria:

* Pregnant or breast-feeding women
* With antecedent or current neurologic disease
* With antecedent or current ophthalmologic disease
* Contraindication for IRMf

Ages: 15 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Volontary subjects : patients suffering from Anorexia Nervosa and control subjects, matched by age and study level
Sampling Method: Non-Probability Sample
Enrollment: 43 (Actual)
Dates: Start 2013-06-07 (Actual); Primary Completion 2020-06-07 (Actual); Study Completion 2020-06-07 (Actual)

PRIMARY OUTCOMES:
Measure of the activation brain areas in self body-recognition network | 15 days
  Level of activation areas in the self body-recognition network measured during fMRI

CONTACTS AND LOCATIONS:
Overall Officials: Olivier Cottencin, MD, PhD, Principal Investigator — University Hospital, Lille
Locations (1):
- CHRU,Hôpital Fontan 2, Lille, France

IPD SHARING:
Plan to Share IPD: No